CLINICAL TRIAL: NCT00371748
Title: TAXUS ATLAS SMALL VESSEL: A Multi-center, Single-arm Study of the TAXUS Liberté™-SR Stent for the Treatment of Patients With de Novo Coronary Artery Lesions in Small Vessels
Brief Title: A Study of the TAXUS Liberté Stent for the Treatment of de Novo Coronary Artery Lesions in Small Vessels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2033; TAXUS ATLAS Small Vessel
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Liberté-SR
- Arm 2 (Other): Historical Comparator: control data derived from a TAXUS V de novo lesion and stent size-matched cohort randomized to receive a single, planned 2.25 mm DES
  Interventions: Device: TAXUS™ Express2
- Arm 3 (Other): Historical Comparator: control data derived from a TAXUS V de novo lesion size-matched cohort randomized to receive a 2.25 mm or 2.5 mm BMS
  Interventions: Device: Express2

INTERVENTIONS:
Device: TAXUS Liberté-SR — Paclitaxel-Eluting Coronary Stent, 2.25 mm
  Arms: Arm 1
Device: TAXUS™ Express2 — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 2
Device: Express2 — Coronary Stent System
  Arms: Arm 3

SUMMARY:
TAXUS ATLAS Small Vessel is a global, multi-center, single-arm, trial of patients with coronary arteries less than 2.5 mm in diameter who are treated with the TAXUS Liberté stent versus an historical TAXUS Express control derived from a subset of lesion-matched TAXUS V patients treated with a 2.25 mm stent. The objective of the study is to evaluate clinical and angiographic outcomes of TAXUS Liberté-SR 2.25 mm stent in de novo lesions. The hypothesis is that the TAXUS Liberté-SR stent has non-inferior safety and efficacy to the TAXUS Express-SR stent in the treatment of de novo lesions in small coronary vessels.

DETAILED DESCRIPTION:
TAXUS ATLAS Small Vessel is a global, multi-center, single-arm, trial of patients receiving the TAXUS Liberté-SR 2.25 mm paclitaxel-eluting stent. The results will be compared with two different historical control groups. The first control group consists of a subset of lesion-matched TAXUS V patients treated with a 2.25 mm TAXUS Express-SR paclitaxel-eluting stent. The objective of this analysis is to evaluate clinical and angiographic outcomes of TAXUS Liberté-SR 2.25 mm stent in de novo lesions versus the TAXUS Express-SR stent. The hypothesis is that the TAXUS Liberté-SR stent has non-inferior safety and efficacy to the TAXUS Express-SR stent in the treatment of de novo lesions in small coronary vessels. The second control group consists of a subset of lesion-matched TAXUS V patients treated with either a 2.5 mm or a 2.25 mm bare metal Express stent. The objective of this analysis is to evaluate clinical and angiographic outcomes of TAXUS Liberté-SR 2.25 mm stent in de novo lesions versus the Express bare metal stent. The hypothesis is that the TAXUS Liberté-SR stent has superior safety and efficacy to the Express bare metal stent in the treatment of de novo lesions in small coronary vessels.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient is at least 18 years old.
2. Eligible for percutaneous coronary intervention (PCI)
3. Documented stable angina pectoris or unstable angina pectoris with documented ischemia, or documented silent ischemia
4. Left ventricular ejection fraction (LVEF) of at least 25%
5. Acceptable candidate for coronary artery bypass grafting (CABG)
6. Patient or legal guardian understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
7. Willing to comply with all specified follow-up evaluations

Angiographic Inclusion Criteria:

1. Only one lesion (target lesion) may be treated with the study stent.However, one additional lesion in a non-target vessel may be treated during the index procedure with a commercially avaiable bare metal stent, heparin-coated stent or TAXUS Express stent.
2. Successful predilation is mandatory for entry into study
3. Target lesion located within a single native coronary artery
4. Target lesion enrolled for treatment may be composed of multiple lesions (not more than 10mm between diseased segments) but must be completely covered by one study stent.
5. Cumulative target lesion length is greater than or equal to 10 mm and less than or equal to 28 mm (visual estimate)
6. Target lesion RVD of 2.25 mm [2.2 - 2.5 mm (visual estimate)]
7. Target lesion diameter stenosis at least 50% (visual estimate)
8. Target lesion is de novo (i.e., a coronary lesion not previously treated)

General Exclusion Criteria:

1. Known hypersensitivity to paclitaxel
2. Any previous, concurrent or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent.
3. Planned use of both the study stent and a non-study stent (i.e., commercial stent) in the treatment of the target vessel
4. Previous or planned treatment with intravascular brachytherapy in the target vessel
5. Planned CABG within 9-months post-index procedure
6. MI within 72 hours prior to the index procedure and/or creatine kinase(CK) >2x the local laboratory's ULN unless CK-MB is <2x ULN
7. Cerebrovascular Accident (CVA) within the past 6 months
8. Cardiogenic Shock
9. Acute or chronic renal dysfunction
10. Contraindication to ASA, or to both clopidogrel and ticlopidine
11. Leukopenia
12. Thrombocytopenia or thrombocytosis
13. Active peptic ulcer or active gastrointestinal (GI) bleeding
14. Known allergy to stainless steel
15. Any prior true anaphylactic reaction to contrast agents
16. Patient is currently, or has been treated with paclitaxel or other chemotherapeutic agents within 12-months of the index procedure
17. Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9-months after the index procedure
18. Male or female with known intention to procreate within 3 months after the index procedure
19. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating
20. Life expectancy of less than 24 months due to other medical condition
21. Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
22. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study

Angiographic Exclusion Criteria:

1. Unprotected and protected left main coronary artery disease (patient with protected left main disease can be enrolled ONLY if the target lesion is in the RCA)
2. Target lesion is ostial in location (within 3.0 mm of vessel origin)
3. Target lesion and/or target vessel proximal to the target lesion is moderately or severely calcified by visual estimate
4. Target lesion and/or target vessel proximal to the target lesion is tortuous
5. Target lesion is located within or distal to a >60 degree bend in the vessel
6. Target lesion involves a bifurcation with a side branch vessel >1.5 mm (visual estimate)
7. Target lesion is totally occluded (TIMI flow <1), either at baseline or predilation
8. Angiographic presence of probable or definite thrombus
9. Pre-treatment of teh target vessel at the index procedure is not allowed with any device except for predilation with balloon angioplasty or cutting balloon
10. A previously treated lesion within the target vessel:

    * <15mm from the target lesion (visual estimate)
    * Performed </= 6 months from index procedure
    * >30% residual stenosis after previous treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percent diameter stenosis - analysis segment at 9 months | 9 Months

SECONDARY OUTCOMES:
Clinical procedural and technical success | 5 Years
Utilization parameters (equipment utilization; catheters, guidewires and balloons, procedure time, fluoroscopic time and amount of contrast used) | 9 months
MACE rates at discharge, 1, 4 and 9 months and 1, 2, 3, 4, and 5 years post-index procedure. | 5 years
Stent thrombosis rate | 5 Years
Target Vessel Failure (TVF) | 5 Years
Target Vessel Revascularization (TVR) | 5 Years
QCA parameters (binary restenosis rate, in-stent %DS, MLD and late loss) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Turco, MD, Principal Investigator — Washington Adventist Hospital; John A Ormiston, MD, Principal Investigator — Mercy Hospital; Peter Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (25):
- United States (19):
  - Mercy General Hospital, Sacramento, California
  - Christiana Hospital, Newark, Delaware
  - Florida Hospital, Orlando, Florida
  - St. John's Hospital, Springfield, Illinois
  - The Heart Center, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Columbia University Medical Center, New York, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - North Ohio Research Elyria Memorial Hospital, Elyria, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - The Pennsylvania State University Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Methodist DeBakey Heart Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
- New Zealand (4):
  - Mercy Angiography Unit, 98 Mountain Road, First Floor, Auckland, Epsom
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore

REFERENCES:
- [Derived] Ormiston JA, Charles O, Mann T, Hall JJ, McGarry T, Cannon LA, Webster MW, Mishkel GJ, Underwood PL, Dawkins KD. Final 5-year results of the TAXUS ATLAS, TAXUS ATLAS Small Vessel, and TAXUS ATLAS Long Lesion clinical trials of the TAXUS Liberte paclitaxel-eluting stent in de-novo coronary artery lesions. Coron Artery Dis. 2013 Jan;24(1):61-8. doi: 10.1097/MCA.0b013e32835b3932. PMID 23232250
- [Derived] Doi H, Maehara A, Mintz GS, Yu A, Wang H, Mandinov L, Popma JJ, Ellis SG, Grube E, Dawkins KD, Weissman NJ, Turco MA, Ormiston JA, Stone GW. Impact of post-intervention minimal stent area on 9-month follow-up patency of paclitaxel-eluting stents: an integrated intravascular ultrasound analysis from the TAXUS IV, V, and VI and TAXUS ATLAS Workhorse, Long Lesion, and Direct Stent Trials. JACC Cardiovasc Interv. 2009 Dec;2(12):1269-75. doi: 10.1016/j.jcin.2009.10.005. PMID 20129555
- [Derived] Mahmud E, Ormiston JA, Turco MA, Popma JJ, Weissman NJ, O'Shaughnessy CD, Mann T, Hall JJ, McGarry TF, Cannon LA, Webster MW, Mandinov L, Baim DS. TAXUS Liberte attenuates the risk of restenosis in patients with medically treated diabetes mellitus: results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2009 Mar;2(3):240-52. doi: 10.1016/j.jcin.2008.12.009. PMID 19463432
- [Derived] Turco MA, Ormiston JA, Popma JJ, Hall JJ, Mann T, Cannon LA, Webster MW, Mishkel GJ, O'Shaughnessy CD, McGarry TF, Mandinov L, Dawkins KD, Baim DS. Reduced risk of restenosis in small vessels and reduced risk of myocardial infarction in long lesions with the new thin-strut TAXUS Liberte stent: 1-year results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2008 Dec;1(6):699-709. doi: 10.1016/j.jcin.2008.09.007. PMID 19463387